CLINICAL TRIAL: NCT01575717
Title: The Effect of Vitamin D Repletion in Patients With Hepatocellular Carcinoma on the Orthotopic Liver Transplant List
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Andrea Branch (Other)
Responsible Party: Sponsor-Investigator, Andrea Branch, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 11-1149; IF# 1333386; HS#: 11-02021
Record Dates: First submitted 2012-04-09; First posted 2012-04-11 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Vitamin D Deficiency; Hepatocellular Carcinoma
Keywords: Vitamin D; hepatocellular carcinoma; liver neoplasms; liver transplantation
MeSH Terms: conditions — Vitamin D Deficiency; Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vitamin D 4000 (Experimental): Subjects taking 4000 IU of vitamin D
  Interventions: Drug: Vitamin D3 4000 IU
- Vitamin D 2000 (Experimental): Subjects taking 2000IU of vitamin D
  Interventions: Drug: Vitamin D3 2000 IU
- No Intervention (No Intervention)

INTERVENTIONS:
Drug: Vitamin D3 4000 IU — Participants with serum 25-hydroxyvitamin D levels of less than or equal to 15ng/ml will take 4000 IU of vitamin D3 daily by mouth for 6 months
  Other Names: Vitamin D 4000
  Arms: Vitamin D 4000
Drug: Vitamin D3 2000 IU — Participants with serum 25-hydroxyvitamin D levels of greater than 15 ng/ml and less than or equal to 25ng/ml will take 2000 IU of vitamin D3 daily by mouth for 6 months
  Other Names: Vitamin D 2000
  Arms: Vitamin D 2000

SUMMARY:
The purpose of this study is to investigate the effect of two different doses of vitamin D3 (2000 IU vs. 4000 IU) on serum 25-hydroxyvitamin D (25OHD) levels in patients with hepatocellular carcinoma on the liver transplant list. The study will help determine the dose of vitamin D3 that is required for patients with liver cancer to reach a normal level of 25OHD in the blood.

DETAILED DESCRIPTION:
Potential participants will be identified from Mount Sinai Hospital's active liver transplant list. The hepatologists at Mount Sinai's Transplant Institute will ask each potential participant if she/he is interested in participating. If the patient expresses an interest in the study, one of the researchers will meet with the patient when the patient is at Mount Sinai for a regular appointment and will describe the study to the potential participant. If a patient continues to be interested in participating, she/he will be given a copy of the IRB-approved consent document to read. The consent document will be used as a guide for explaining the study in detail to the patient. If the patient's preferred language is Spanish, she/he will be given a consent document in Spanish and the study will be explained in Spanish.

Once the subject's 25(OH)D level is known, if the subject's 25(OH)D level is ≤ 15 ng/ml, the participant will be contacted by one of the investigators on the research team and instructed to begin taking 2 tablets per day (4000 IU total) of vitamin D. If the subject's 25(OH)D level is greater than 15 and ≤ 25, the participant will be contacted by one of the investigators on the research team and told to begin taking 1 tablet (2000 IU total) per day of vitamin D. If the participant's vitamin D level is < 25 ng/ml, they are considered Vitamin D insufficient/deficient. If the Serum Vitamin D is > 25 ng/ml they will be informed that they are not to take any vitamin D and they will be followed as controls for this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and older)
* Diagnosis of hepatocellular carcinoma
* On the list awaiting liver transplantation
* Able to give informed consent
* Expected to receive care following liver transplantation at the Mount Sinai School of Medicine
* Any race/ethnicity/socioeconomic status

Exclusion Criteria:

* Pediatric patient (less than 18 years of age)
* Unable to give informed consent
* Untreated primary hyperparathyroidism (ICD9 codes 252.01XX and 252.00XX)
* Untreated hypercalcemia (serum calcium level > 11 mg/dl; ICD9 codes 275.42XX, 259.3XX, 252.00F)
* Pregnancy (will be determined by asking the patient and reviewing the medical record)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Change in serum levels of 25-hydroxyvitamin D | at baseline, and at 3 and 6 months
  Change in serum levels of 25-hydroxyvitamin D at 3 months and 6 months compared to baseline

SECONDARY OUTCOMES:
Change in serum levels of liver enzymes (ALT, AST and Alk phos) | at baseline, and at 3 and 6 months
  Change in serum levels of liver enzymes (ALT, AST and Alk phos) at 3 months and at 6 months compared to baseline
Change in serum creatinine | at baseline, and at 3 and 6 months
  Change in serum creatinine at 3 months and at 6 months compared to baseline
Serum Calcium | at 3 months
Serum Calcium | at 6 months
Change in coagulation profile (PT/PTT and INR) | at baseline, and at 3 and 6 months
  Change in coagulation profile (PT/PTT and INR) at 3 months and at 6 months compared to baseline
Change in Model for End stage Liver Disease score (MELD) | at baseline, and at 3 and 6 months
  Change in Model for End stage Liver Disease score (MELD) at 3 months and at 6 months compared to baseline.
  Calculated using the following formula: Meld = 10x ((0.957 x Ln(creatinine mg/dl)) + (0.378 x Ln(bilirubin mg/dl)) + (1.120 x Ln(INR)) + 0.643)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea D Branch, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- The Mount Sinai Hospital, New York, New York, United States

REFERENCES:
- [Background] Malham M, Jorgensen SP, Ott P, Agnholt J, Vilstrup H, Borre M, Dahlerup JF. Vitamin D deficiency in cirrhosis relates to liver dysfunction rather than aetiology. World J Gastroenterol. 2011 Feb 21;17(7):922-5. doi: 10.3748/wjg.v17.i7.922. PMID 21412501
- [Background] Wibaux C, Legroux-Gerot I, Dharancy S, Boleslawski E, Declerck N, Canva V, Mathurin P, Pruvot FR, Cortet B. Assessing bone status in patients awaiting liver transplantation. Joint Bone Spine. 2011 Jul;78(4):387-91. doi: 10.1016/j.jbspin.2011.03.001. Epub 2011 May 11. PMID 21565541
- [Background] Arteh J, Narra S, Nair S. Prevalence of vitamin D deficiency in chronic liver disease. Dig Dis Sci. 2010 Sep;55(9):2624-8. doi: 10.1007/s10620-009-1069-9. Epub 2009 Dec 4. PMID 19960254
- [Background] Ninkovic M, Love SA, Tom B, Alexander GJ, Compston JE. High prevalence of osteoporosis in patients with chronic liver disease prior to liver transplantation. Calcif Tissue Int. 2001 Dec;69(6):321-6. doi: 10.1007/s00223-001-2028-4. PMID 11800228
- [Background] Loria I, Albanese C, Giusto M, Galtieri PA, Giannelli V, Lucidi C, Di Menna S, Pirazzi C, Corradini SG, Mennini G, Rossi M, Berloco P, Merli M. Bone disorders in patients with chronic liver disease awaiting liver transplantation. Transplant Proc. 2010 May;42(4):1191-3. doi: 10.1016/j.transproceed.2010.03.096. PMID 20534258
- [Background] Bitetto D, Fabris C, Falleti E, Fornasiere E, Fumolo E, Fontanini E, Cussigh A, Occhino G, Baccarani U, Pirisi M, Toniutto P. Vitamin D and the risk of acute allograft rejection following human liver transplantation. Liver Int. 2010 Mar;30(3):417-44. doi: 10.1111/j.1478-3231.2009.02154.x. Epub 2009 Oct 22. PMID 19849776